CLINICAL TRIAL: NCT02101424
Title: Monitoring of Overdose Patients With and Without Supplemental Oxygen in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 10-3179
Record Dates: First submitted 2013-10-24; First posted 2014-04-02 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Overdose
Keywords: Overdose; Emergency Department; Supplemental Oxygen; Pulse Oximeter; Capnography
MeSH Terms: conditions — Drug Overdose; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Overdose

SUMMARY:
This study will compare the data from pulse oximeters to capnographers as they are used to monitor patients who are being observed in the Emergency Department for a suspected overdose of alcohol or other drugs. The investigators will compare monitor data from patients who are and are not on supplemental oxygen, the ability of the monitors to predict the occurrence of airway interventions, and to detect ventilator changes noted on the opposing monitor. There will not be any interventions during this study other than the collection of data from the monitors and observation of the care of patients.

ELIGIBILITY:
Inclusion Criteria:

* Airway is being monitored as a result of overdose

Exclusion Criteria:

* Under 18 years old
* Unable to give informed consent at baseline
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department at an urban county hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Airway Interventions Performed by ED Staff | 4 hours
  Addition or increase in supplemental oxygen, stimulation to induce respiration, airway repositioning, bag-valve-mask application, positive pressure ventilation, intubation, airway suctioning, vomiting, medication administration, transfer to a higher level of care.
Pulse oximetry | 4 hours
  recorded every 5 minutes and at the time of clinical interventions
End tidal CO2 | 4 hours
  recorded every 5 minutes and at the time of any clinical intervention

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States